CLINICAL TRIAL: NCT03464383
Title: Anxiety and Depression in Epilepsy: A Pilot Epileptologist-Driven Treatment Study
Brief Title: Anxiety and Depression in Epilepsy: A Treatment Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00048584; 5UL1TR001420-03 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-09

CONDITIONS: Anxiety; Depression; Epilepsy
Keywords: Neurologic Disorders; Chronic Care; Management; Treatment; SSRI Medication; SNRI Medication; Learning Healthcare System
MeSH Terms: conditions — Anxiety Disorders; Depression; Epilepsy; Nervous System Diseases | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups. Those randomized to the intervention group will receive an epileptologist-driven medication treatment for anxiety and depression, carried out directly in the epilepsy clinic during a regularly scheduled visit and supported by advanced practice provider (APP). Those randomized to the control group will receive an referral order to psychiatry placed by their epileptologist.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment phone calls for gathering scaled instrument scores will be carried out by a second study coordinator, blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Epileptologist-Driven Treatment (Experimental): The intervention will consist of initiating a chronic care management plan in the epilepsy clinic and an initial prescription from the epileptologist for escitalopram 10mg daily. Escitalopram dose adjustment will be made based on biweekly repeated screening of anxiety and depression symptoms, as well as side effects identified on biweekly telephone calls or the 6-week advanced practice provider (APP) follow up visit. Escitalopram dose may be titrated up to a maximum of 20mg daily in 5-10mg increments every 2 weeks for treatment effect, or titrated down to 5mg if needed for adverse effects. If a participant is unable to tolerate escitalopram, then venlafaxine XR 37.5mg will be substituted, to be titrated in a similar manner biweekly based on side effects and anxiety and depression symptoms (with 37.5-75mg increment dose changes and maximum dose of 225mg daily).
  Interventions: Drug: Escitalopram 10mg
- Standard of Care (Active Comparator): A psychiatry referral order placed by epileptologist under typical care circumstances (internal or external referral based on the participant's geographic preferences). Internal referrals will be processed by current clinic/institutional protocols. External referral orders will be printed and provided to the patient along with brief instructions on how to find a provider covered by the patient's insurance.
  Interventions: Other: Referral to Psychiatry
- Survey Arm (Other): This option will be offered to individuals who are found to have anxiety or depression symptoms on screening but who are found to be ineligible for intervention arms of the study, or those who are eligible for the intervention arm but decline to participate in the intervention.
  Interventions: Other: Survey only

INTERVENTIONS:
Drug: Escitalopram 10mg — Participants will be given escitalopram 10mg by mouth daily and will be followed up with at 2, 4, 6, 8, and 10 weeks. Medication will be adjusted if side effects occur. If unable to tolerate escitalopram, then venlafaxine XR (Effexor XR) 37.5mg will be substituted.
  Other Names: Lexapro
  Arms: Epileptologist-Driven Treatment
Other: Referral to Psychiatry — Participants randomized to control will have a psychiatry referral order placed by the treating epileptologist under typical care circumstances. This will be an internal or external referral order based on patient preference. If external, the order will be printed along with instructions for the patient to follow to find a provider covered by insurance.
  Arms: Standard of Care
Other: Survey only — One time survey will be offered to individuals who are found to have anxiety or depression symptoms on screening but who are ineligible for the treatment component of the study, or who decline the treatment study.
  Arms: Survey Arm

SUMMARY:
As a potential solution to address high rates of depression and anxiety seen in epilepsy patients and poor mental health care access, this randomized trial aims to study treatment for anxiety and depression in epilepsy taking place directly within the epilepsy clinic vs. psychiatry referral (typical care). Patients that meet eligibility criteria, including significant symptoms of depression and/or anxiety, will be randomized to the either the intervention group or the control group. Patients that do not meet eligibility requirement or decline the study intervention will have the option of participating in the survey arm of the study. The intervention will consist of an initial prescription for an FDA-approved medication to treat depression/anxiety and telephone-based chronic care management plan for repeated symptom measurement and side effect surveillance. The control group will receive usual care, which is a referral order to psychiatry placed by their treating neurologist. Participants in the survey arm of the study will complete a one time survey.

DETAILED DESCRIPTION:
This trial is an innovative learning healthcare system approach to translate the concept of measurement-based depression care into a specialty clinic setting and extend the concept to treat depression and/or anxiety. The investigators' neurologist/APP-administered medication intervention utilizes FDA-approved drugs with advantageous features for use in epilepsy (escitalopram and venlafaxine) and a telephone-based chronic care management plan for repeated symptom measurement and side effect surveillance. The proposed intervention may overcome barriers to implementing mental health treatment interventions in generalized clinical settings by using healthcare providers commonly present in specialty clinics (physicians and APPs) along with a billable, best practices chronic care management intervention package and EMR-based clinical tools.To test this idea, the investigators seek to pilot a randomized trial of neurologist/APP medication management of depression and anxiety versus usual care with psychiatry referral in the epilepsy clinic, using epilepsy as a paradigm for chronic medical illness with high prevalence of psychiatric comorbidity. The optional survey arm is to help investigators understand the population that do not meet criteria or refuse intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 18 or older
* Ability to take oral medication and the willing to adhere to the intervention regimen
* Minimum of 1 prior clinic visit at the Comprehensive Epilepsy Center
* Ability to complete questionnaires independently
* Diagnosis of epilepsy: EEG with documented seizure or epileptiform discharges OR non-epileptiform EEG and seizure remission with antiseizure drug OR treating epileptologist's leading clinical impression is epilepsy
* (Neurological Disorders Depression Inventory for epilepsy, NDDI-E score greater than 15 and/or Generalized Anxiety Disorder-7, GAD-7 score greater than or equal to 10

Exclusion Criteria:

* Pregnancy or lactation
* Known allergic reactions to escitalopram or venlafaxine
* Comorbid psychogenic nonepileptic seizures
* Prior psychiatric hospitalization
* Prior suicide attempt
* History of manic or psychotic symptoms (past manic episode (SCID-I), or psychotic symptom screen positive)
* Current treatment by a psychiatrist or counselor/therapist
* Active suicidality at the time of screening
* Current treatment with buspirone or an SSRI/SNRI/atypical antidepressant (specifically bupropion, fluoxetine, levomilnacipran, citalopram, milnacipran, desvenlafaxine, mirtazapine, duloxetine, paroxetine, escitalopram, sertraline, fluvoxamine, venlafaxine, vilazodone, vortioxetine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Munger Clary, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Epileptologist-Driven Treatment: The intervention will consist of initiating a chronic care management plan in the epilepsy clinic and an initial prescription from the epileptologist for escitalopram 10mg daily. Escitalopram dose may be titrated up to a maximum of 20mg daily in 5-10mg increments every 2 weeks for treatment effect, or titrated down to 5mg if needed for adverse effects. If a participant is unable to tolerate escitalopram, then venlafaxine XR 37.5mg will be substituted, to be titrated in a similar manner biweekly based on side effects and anxiety and depression symptoms (with 37.5-75mg increment dose changes and maximum dose of 225mg daily).
Period: Overall Study
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Started | 3 | 3 | 63
Completed | 2 | 2 | 63
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm | Total
Number analyzed (Participants) | 3 | 3 | 63 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 61 | 67
  >=65 years | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (6.1) | 41.3 (4.0) | 42.2 (13.5) | 42.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 40 | 42
  Male | 2 | 2 | 23 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 3 | 47 | 53
  Unknown or Not Reported | 0 | 0 | 12 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 9 | 10
  White | 3 | 2 | 48 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 63 | 69

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Intervention
Description: Percentage of participants who report taking the prescribed medication at 12 weeks and who have completed at least 2 of the chronic care management scheduled visits (telephone or clinic visit)
Time Frame: 12 weeks
Population: This outcome only pertains to the experimental arm. This was an intention-to treat analysis including all who were randomized to the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Number analyzed (Participants) | 3 | 0 | 0
Participants | 2 | 0 | 0

2. Secondary Outcome: Accrual
Description: Percentage of patients screened for the trial who are eligible
Time Frame: baseline
Population: Number of participants analyzed were not all consented or randomized. These were pre-screening numbers.
Measure: Count of Participants; unit: Participants
Groups:
- Epileptologist-Driven Treatment Plus Standard of Care Arm: Combined treatment arms
Arm/Group | Epileptologist-Driven Treatment Plus Standard of Care Arm
Number analyzed (Participants) | 681
Participants | 19

3. Secondary Outcome: Participants Eligible for Consent Into Treatment Arms
Description: Percent eligible who consent to participate in treatment study
Time Frame: baseline
Population: This is the number who were pre-screened and who were eligible to consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Epileptologist-Driven Treatment Plus Standard of Care Arm
Number analyzed (Participants) | 19
Participants | 6

4. Secondary Outcome: Retention
Description: Percentage of participants who complete the 12 week outcome assessment
Time Frame: 12 weeks
Population: This was an intention-to treat analysis including all who were randomized to the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Number analyzed (Participants) | 3 | 3 | 0
Participants | 2 | 2 | 0

5. Secondary Outcome: Efficacy - Depression Symptoms
Description: Using Beck Depression Inventory-II (BDI-II) among those with high depression at baseline. The BDI-II is a self-report measure of depressive symptoms. Scores range from 0 to 63, with a higher score representing higher levels of depressive symptoms and higher scores representing worse outcome.
Time Frame: baseline
Population: This outcome does not apply to survey arm. Baseline measurements were done before subjects in each treatment arm were lost to follow up and withdrew consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Number analyzed (Participants) | 3 | 3 | 0
score on a scale | 26.7 (3.5) | 21.0 (7.2) |

6. Secondary Outcome: Efficacy - Depression Symptoms
Description: Beck Depression Inventory-II (BDI-II) among those with high depression at baseline. The BDI-II is a self-report measure of depressive symptoms. Scores range from 0 to 63, with a higher score representing higher levels of depressive symptoms and higher scores representing worse outcome.
Time Frame: 12 weeks
Population: This outcome does not apply to survey arm. 12 week measurements were done after subjects in each treatment arm were lost to follow up and withdrew consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Number analyzed (Participants) | 2 | 2 | 0
score on a scale | 25.0 (5.7) | 17.0 (8.5) |

7. Secondary Outcome: Efficacy - Anxiety Symptoms
Description: Beck Anxiety Index (BAI) among those with high anxiety at baseline. The BAI is a self-report measure used for measuring the severity of anxiety. Scores range from 0 to 63, with a higher score representing more severe anxiety symptoms and higher scores representing worse outcomes.
Time Frame: baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Number analyzed (Participants) | 3 | 3 | 0
score on a scale | 18.0 (9.6) | 10.5 (2.1) |

8. Secondary Outcome: Efficacy - Anxiety Symptoms
Description: as for outcome 7
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
Number analyzed (Participants) | 2 | 1 | 0
score on a scale | 9.5 (9.2) | 11 |

ADVERSE EVENTS:
Time Frame: Baseline through 12 weeks for experimental and standard of care arms. For survey arm, from survey completion to time when incentive gift card communications were completed.
Arm/Group | Epileptologist-Driven Treatment | Standard of Care | Survey Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/63
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/63
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epileptologist-Driven Treatment (N=3) | Standard of Care (N=3) | Survey Arm (N=63)
sudden unexpected death in epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epileptologist-Driven Treatment (N=3) | Standard of Care (N=3) | Survey Arm (N=63)
tooth pain from impacted wisdom tooth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
night sweats (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03464383/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03464383/Prot_SAP_001.pdf